CLINICAL TRIAL: NCT06099782
Title: A Phase 2 Study to Evaluate Patient Reported Preference for Subcutaneous Pembrolizumab Coformulated With Hyaluronidase (MK-3475A) Over Intravenous Pembrolizumab Formulation in Participants With Multiple Tumor Types (MK-3475A-F11)
Brief Title: A Study of Participant Reported Preference for Subcutaneous Pembrolizumab Coformulated With Berahyaluronidase Alfa (MK-3475A) Over Intravenous Pembrolizumab (MK-3475) Formulation in Multiple Tumor Types (MK-3475A-F11)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3475A-F11; 2023-506017-22 (Registry Identifier: EU CT); U1111-1293-0814 (Registry Identifier: UTN); MK-3475A-F11 (Other: MSD); jRCT2051230147 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer; Renal Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pembrolizumab (+) Berahyaluronidase alfa SC →Pembrolizumab IV (Experimental): In the treatment crossover period, participants will receive pembrolizumab (+) berahyaluronidase alfa SC followed by pembrolizumab IV. After completion of the treatment crossover period, participants will enter the treatment continuation period, where they will receive their preferred intervention for up to ~1 year for renal cell carcinoma (RCC) and melanoma and for up to ~2 years for non-small cell lung cancer (NSCLC).
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Biological: Pembrolizumab
- Arm B: Pembrolizumab IV→pembrolizumab (+) berahyaluronidase alfa SC (Active Comparator): In the treatment crossover period, participants will receive pembrolizumab IV followed by pembrolizumab (+) berahyaluronidase alfa SC. After completion of the treatment crossover period, participants will enter the treatment continuation period, where they will receive their preferred intervention for up to ~1 year for RCC and melanoma and for up to ~2 years for NSCLC.
  Interventions: Biological: Pembrolizumab (+) Berahyaluronidase alfa; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab (+) Berahyaluronidase alfa — Fixed dose coformulated product of hyaluronidase/pembrolizumab adminstered via SC injection.
  Other Names: MK-3475A
Biological: Pembrolizumab — Administered via IV infusion
  Other Names: MK-3475, KEYTRUDA®

SUMMARY:
The purpose of this study is to evaluate participant preference for coformulated hyaluronidase/pembrolizumab pembrolizumab (+) berahyaluronidase alfa administered subcutaneously (SC) over pembrolizumab (MK-3475) administered intravenously (IV) in participants with multiple tumor types. There will be no hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed early stage or advanced/ metastatic solid tumor by pathology report and meet the following conditions based on tumor type:

  * Surgically resected Stage IIB and IIC (pathological or clinical), or III cutaneous melanoma per American Joint Committee on Cancer (AJCC) eighth edition.
  * Surgically resected renal cell carcinoma (RCC) with intermediate-high or high risk of recurrence as defined by the Fuhrman grading status.
  * Stage IV non-small cell lung cancer (NSCLC) per AJCC eight edition, with an anti-programmed cell death ligand 1 (PD-L1) tumor proportion score (TPS) ≥50% determined using the Dako PD-L1 immunohistochemistry (IHC) 22C3 pharmDx diagnostic kit, and confirmation that epidermal growth factor receptor (EGFR-), anaplastic lymphoma kinase (ALK-), or c-ros oncogene 1 (ROS1)- directed therapy is not indicated as primary therapy.
* Has a life expectancy of at least 3 months.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART).
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load before randomization.
* Participants with history of hepatitis C virus (HCV) infection are eligible if have completed curative antiviral therapy at least 4 weeks before randomization and HCV viral load is undetectable at screening.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 3 days before the start of study intervention.

Exclusion Criteria:

* Non-small cell lung cancer (NSCLC) participants with a diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements.
* Melanoma participants with ocular, mucosal, or conjunctival melanoma.
* Renal Cell Carcinoma (RCC) participants who have had major surgery, other than nephrectomy, within 12 weeks before randomization.
* Has received prior radiotherapy for RCC.
* RCC participants who have residual thrombus post nephrectomy in the vena renalis or vena cava.
* Has received prior therapy with an anti-programmed cell death 1 protein (PD-1), PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids.
* Received prior systemic anticancer therapy for their metastatic NSCLC. Note: Prior treatment with neoadjuvant or adjuvant therapy for nonmetastatic NSCLC is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC.
* Received radiation therapy to the lung that is >30 Gray within 6 months of start of study intervention.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Has diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication.
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has active infection requiring systemic therapy.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Has history of allogeneic tissue/solid organ transplant corticosteroids.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has not adequately recovered from major surgery or have ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Prefer Pembrolizumab (+) Berahyaluronidase alfa Subcutaneous (SC) on Patient Preference Questionnaire (PPQ) Question 1 | ~Day 106
  The PPQ is an instrument that has been developed from participant interviews and includes questions to evaluate directly from participants their preference regarding mode of administration, as well as the strength of the preference, and the reason for the preference. Question 1 in PPQ evaluates participants' preferred method of administration with response options of IV, SC or no preference. The percentage of participants who prefer SC will be reported.

SECONDARY OUTCOMES:
Percentage of Responses From Participants to the Two Main Reasons for Their Preferred Method of Administration as Assessed on PPQ Question 3 | ~Day 106
  The PPQ is an instrument that has been developed from patient interviews and includes questions to evaluate directly from participants their preference regarding mode of administration, as well as the strength of the preference, and the reason for the preference. Question 3 in PPQ evaluates two main reasons for participants' preference for one of the administration methods with response options of feels less emotionally distressing, requires less time in the clinic, lower level injection-site pain, among others. The percentage of responses from participants to the two main reasons for their preferred method of administration, as assessed on PPQ Question 3 will be reported.
Percentage of Participants by Their Level of Satisfaction With the SC Method of Administration as assessed on Therapy Administration Satisfaction Questionnaire - Subcutaneous (TASQ-SC) Question 1 | Up to ~Day 106
  The TASQ SC is a 12-item questionnaire that asks questions regarding different aspects of participants' satisfaction with SC administration, experiences related to administration, convenience, time. Question 1 in TASQ SC evaluates participants' satisfaction or dissatisfaction with SC administration. The percentage of participants by their level of satisfaction with the SC method of administration as assessed on TASQ-SC Question 1 will be reported.
Percentage of Participants by Their Level of Satisfaction With the IV Method of Administration as assessed on Therapy Administration Satisfaction Questionnaire -Intravenous (TASQ-IV) Question 1 | Up to ~Day 106
  The TASQ IV is a 12-item questionnaire that asks questions regarding different aspects of participants' satisfaction with IV administration, experiences related to administration, convenience, time. Question 1 in TASQ IV evaluates participants' satisfaction or dissatisfaction with IV administration. The percentage of participants by their level of satisfaction with the IV method of administration as assessed on TASQ-IV Question 1 will be reported.
Percentage of Participants Who Choose Pembrolizumab (+) Berahyaluronidase alfa SC for the Study Treatment Continuation Period | ~Day 106
  The percentage of participants who choose SC treatment for the continuation period in the study will be reported.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study drug due to an AE | Up to ~24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (45):
- United States (8):
  - Russell Medical ( Site 0160), Alexander City, Alabama
  - Alaska Oncology and Hematology ( Site 0121), Anchorage, Alaska
  - Highlands Oncology Group-Research Department ( Site 0133), Springdale, Arkansas
  - Marin Cancer Care ( Site 0148), Greenbrae, California
  - Holy Cross Hospital-Clinical Research ( Site 0159), Fort Lauderdale, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0113), Orange City, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 0112), Marietta, Georgia
  - Kadlec Clinic Hematology and Oncology ( Site 0103), Kennewick, Washington
- Argentina (3):
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0300), Mar del Plata, Buenos Aires
  - Fundación Respirar ( Site 0302), Buenos Aires, Buenos Aires F.D.
  - Instituto San Marcos ( Site 0305), San Juan
- Australia (2):
  - Port Macquarie - Mid North Coast Cancer Institute-Medical Oncology ( Site 1001), Port Macquarie, New South Wales
  - Frankston Hospital-Oncology and Haematology ( Site 1007), Frankston, Victoria
- Chile (7):
  - Clínica Puerto Montt ( Site 0404), Port Montt, Los Lagos Region
  - FALP-UIDO ( Site 0401), Santiago, Region M. de Santiago
  - Oncovida ( Site 0403), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Hemato-Oncology ( Site 0407), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0402), Santiago, Region M. de Santiago
  - Centro Investigacion Cancer James Lind ( Site 0408), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0400), Viña del Mar, Región de Valparaíso
- France (5):
  - CENTRE LEON BERARD-onco dermatology ( Site 0600), Lyon Cedex08, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire de Caen Normandie-DERMATOLOGY ( Site 0604), Caen, Calvados
  - Clinique Francois Chenieux ( Site 0603), Limoges, Haute-Vienne
  - HIA Sainte Anne-Pneumology ( Site 0601), Toulon, Var
  - Hôpital Bichat - Claude-Bernard ( Site 0605), Paris, Île-de-France Region
- Japan (2):
  - Bell Land General Hospital ( Site 1101), Sakai, Osaka
  - Tokyo Women's Medical University ( Site 1100), Tokyo
- New Zealand (2):
  - Auckland City Hospital-Cancer & Blood Research ( Site 1051), Auckland
  - Bowen Hospital ( Site 1050), Wellington
- Poland (4):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 0701), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier, Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0702), Koszalin, West Pomeranian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 0703), Szczecin, West Pomeranian Voivodeship
- South Africa (8):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 0808), Port Elizabeth, Eastern Cape
  - Medical Oncology Centre of Rosebank ( Site 0805), Johannesburg, Gauteng
  - Nosworthy Oncology ( Site 0807), Johannesburg, Gauteng
  - Steve Biko Academic Hospital-Medical Oncology ( Site 0804), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 0800), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 0801), Sandton, Gauteng
  - Cape Town Oncology Trials ( Site 0802), Cape Town, Western Cape
  - CANCERCARE RONDEBOSCH ONCOLOGY-Cancercare Rondebosch Oncology ( Site 0806), Cape Town, Western Cape
- Turkey (Türkiye) (4):
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 0903), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0900), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 0901), Ankara
  - Ege Universitesi Hastanesi ( Site 0902), Izmir

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26236&tenant=MT_MSD_9011